CLINICAL TRIAL: NCT06809504
Title: Restoring Functionality: Occupational Therapy Interventions in Substance Use Drug Rehabilitation
Brief Title: To Assess the Effectiveness of Structured Occupational Therapy (OT) Interventions on Patients With SUD in Inpatient Department (IPD) Settings, Focusing on Improvements in Cognitive, Physical, and Functional Domains
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hammad Mursaleen (Other)
Responsible Party: Sponsor-Investigator, Hammad Mursaleen, Mr, Foundation of Medical Research and Laboratories, Pakistan
Organization: Foundation of Medical Research and Laboratories, Pakistan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMRL01; FMRL01 (Other: Foundation of medical research and laboratory)
Record Dates: First submitted 2025-01-28; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Substance Abuse Disorder
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: 12 sessions over 4 weeks, 45-minute sessions divided into:
  * 15 minutes for physical exercises
  * 15 minutes for psychoeducation
  * 15 minutes for cognitive tasks and routine planning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Exercise based intervention was given for 12 sessions over 4 weeks, 45-minute sessions
  Interventions: Behavioral: Exercise based intervention

INTERVENTIONS:
Behavioral: Exercise based intervention — 12 sessions over 4 weeks, 45-minute sessions divided into:
  o 15 minutes for physical exercises

SUMMARY:
OT emphasis lies within the scope of improving daily life activities, cognitive and physical performance in order to regain the proper social role. This work assesses the impact of a 12 session structured OT intervention program for patients with SUD in IPD. Benefitting from checklists like the Montreal Cognitive Assessment (MoCA), the Barthel Index, the Lawton-Brody IADLs scale, it substantiates attaining enhancements in expressive cognitive functions, ADLs, and IADLs to understand how selected OT intervention modalities can enhance functional capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Substance abused disorder
* Admitted in rehabilitation center

Exclusion Criteria:

* Severe cognitive impairment
* Physical disability

Max Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 12 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2024-11-12 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA): | baseline and after 12 weeks of intervention
  The MoCA offers assessment of many cognitive aspects, it presents assessments for attention, memory, language, visual construction, executive functions, and orientation.

CONTACTS AND LOCATIONS:
Locations (1):
- FMRL, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided